CLINICAL TRIAL: NCT02836028
Title: A Phase 2, Multiple-Cohort, Open-Label, International Study of Talazoparib Monotherapy and Talazoparib Plus Temozolomide in Women With Relapsed Ovarian, Fallopian Tube, and Peritoneal Cancer
Brief Title: A Study Evaluating Talazoparib in Relapsed Ovarian, Fallopian Tube, and Peritoneal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Myriad Genetic Laboratories, Inc. (Industry); Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDV3800-11
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — talazoparib; Temozolomide

ARMS (2):
- talazoparib (Experimental): Cohorts 1A (PARP inhibitor naïve), 2A (PARP inhibitor sensitive), and 3A (PARP inhibitor refractory)
  Interventions: Drug: Talazoparib
- talazoparib + temozolomide (Active Comparator): Cohorts 1B (PARP inhibitor naïve), 2B (PARP inhibitor sensitive), and 3B (PARP inhibitor refractory)
  Interventions: Drug: Talazoparib; Drug: Temozolomide

INTERVENTIONS:
Drug: Talazoparib — Talazoparib monotherapy 1mg/day orally
  Other Names: MDV3800; BMN673
Drug: Temozolomide — temozolomide 37.5 mg/m2 on days 1-5 of each cycle
  Arms: talazoparib + temozolomide

SUMMARY:
The purpose of this phase 2, multiple-cohort, randomized, open-label, international study of talazoparib (a poly (ADP-ribose) polymerase (PARP) inhibitor) is to compare the efficacy and safety of talazoparib monotherapy and talazoparib plus temozolomide in women with relapsed ovarian, fallopian tube, and peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of age and willing and able to provide informed consent
* Relapsed, histologically confirmed ovarian, fallopian tube, and peritoneal cancer. Histologic subtypes include serous, endometrioid, clear-cell, mixed, undifferentiated histology, and carcinosarcoma.
* Sufficient archival tumor tissue available or consent to a fresh tissue biopsy for biomarker analysis. Consent to blood sample collection for biomarker analysis is required.
* Disease progression per RECIST 1.1 during or after the last treatment. Have metastatic disease with at least 1 target tumor lesion measurable per RECIST 1.1 on the screening scan. Lesions used for biopsies cannot be designated as a measurable lesion for RECIST 1.1 assessments.
* Additional criteria for cohort 1 include the following:
* Have a deleterious germline or a somatic BRCA1 or BRCA2 mutation, or a high diagnostic HRD test score (myChoice score ≥ 42), which represents a loss of DNA repair function based on testing performed at a sponsor-approved laboratory
* Received at least 1 and no more than 3 platinum-based chemotherapy regimens (prior bevacizumab is allowed) and the last dose is ≥ 28 days before randomization
* No prior PARP inhibitor treatment (COHORT 1 ONLY)
* Additional criteria for cohorts 2 and 3 include the following:
* Received at least 2 platinum-based chemotherapy regimens (including first-line chemotherapy; prior bevacizumab is allowed) and the last dose is ≥ 28 days before randomization
* Received prior PARP inhibitor treatment as a single agent or in combination therapy regimen and the last dose is ≥ 28 days before randomization, as follows:
* For cohort 2 only: Received PARP inhibitor treatment for ≥ 6 months and had a response of CR, PR, or stable disease for ≥ 6 months
* For cohort 3 only: Received PARP inhibitor treatment for < 6 months with no response (disease progression or stable disease)
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Estimated life expectancy of ≥ 3 months.
* Able to swallow drugs, have no known intolerance to study drugs or excipients, and able to comply with study requirements.

Exclusion Criteria:

* Have not recovered (recovery is defined as National Cancer Institute Common Terminology Criteria for Adverse Events [CTCAE] grade ≤ 1) from the acute toxicities of previous therapy, except treatment-related alopecia or laboratory abnormalities otherwise meeting eligibility requirements.
* Use of any investigational agent within 14 days before randomization.
* Had > 2 paracentesis procedures within 28 days before randomization.
* Major surgery within 14 days before randomization.
* Requirement for intravenous alimentation (at the time of randomization).
* Diagnosis of MDS.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Determine Objective Response Rate (ORR) | Anticipated in about 44 months following first patient enrolled

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Anticipated in about 44 months following first patient enrolled
PFS at 24 weeks | Anticipated in about 44 months following first patient enrolled
Gynecologic Cancer Intergroup (GCIG) CA125 response rate | Anticipated in about 44 months following first patient enrolled
Clinical benefit rate at 24 weeks | Anticipated in about 44 months following first patient enrolled
Duration of response (DOR) | Anticipated in about 44 months following first patient enrolled
Time to response | Anticipated in about 44 months following first patient enrolled
Overall survival | Anticipated in about 44 months following first patient enrolled
Safety as assessed by percentage of patients with any Adverse Event (AE), AE leading to Study Drug Discontinuation, AE leading to death, SAE, AE related to study drug, SAE related to study drug. | Anticipated in about 44 months following first patient enrolled
Pharmacokinetics of talazoparib as assessed by trough plasma concentrations | Anticipated in about 44 months following first patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer